CLINICAL TRIAL: NCT06736561
Title: A Multicenter Real-world Clinical Study on the Efficacy and Safety of Ensartinib As Neoadjuvant Treatment for Anaplastic Lymphoma Kinase (ALK) Positive Non-small Cell Lung Cancer (NSCLC) Patients.
Status: Not yet recruiting | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Jianqun Ma, archiater, Harbin Medical University
Other Study IDs: 2024-275-IIT
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: ALK Positive; Ensartinib; NSCLC; Neoadjuvant Therapy
Keywords: ALK Positive; Ensartinib; NSCLC; Neoadjuvant therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Data on the efficacy and safety of patients who had previously used enshatinib in the neoadjuvant phase were retrospectively collected
- Cohort 2: Akl-positive patients received enshatinib monotherapy neoadjuvant therapy for 6-12 weeks
- Cohort 3: Alk-positive patients received neoadjuvant therapy that included enshatinib and did not meet cohort 2 inclusion criteria

SUMMARY:
Explore the efficacy and safety of Ensartinib in neoadjuvant treatment for ALK-positive non-small cell lung cancer in the real world.This is a real-world study of patients receiving enshatinib-based neoadjuvant therapy with R0 resection, divided into retrospective cohort 1, prospective cohort 2, and prospective cohort 3. The dose, duration, and whether to combine or sequentially treat enshatinib were clinical decisions made by the investigator on a patient-specific basis.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1: Female or male aged >=18 years;
2. Cohort 1: Received neoadjuvant treatment with Ensartinib before the project started;
3. Cohort 1: Diagnosed with clinical stage II-III resectable or potentially resectable (T1-4 N2 M0) ALK-positive NSCLC before neoadjuvant treatment;
4. Cohort 1: Confirmed ALK positive by immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), next-generation sequencing (NGS), or other non-specific sequencing methods before receiving ALK inhibitor therapy.
5. Cohort 2: Female or male aged >=18 years;
6. Cohort 2: Intended to receive Ensartinib monotherapy as neoadjuvant treatment for 6-12 weeks;
7. Cohort 2: Diagnosed with clinical stage II-III resectable or potentially resectable (T1-4 N2 M0) ALK-positive NSCLC before neoadjuvant treatment;
8. Cohort 2: Confirmed ALK positive by immunohistochemistry (IFL), fluorescence in situ hybridization (FISH), next-generation sequencing (NGS), or other non-specific sequencing methods before receiving ALK inhibitor therapy;
9. Cohort 2: Signed informed consent form;
10. Cohort 3: Female or male aged >=18 years;
11. Cohort 3: Intended to receive neoadjuvant treatment including Ensartinib, but not meeting the inclusion criteria for Cohort 2;
12. Cohort 3: Diagnosed with clinical stage II-III resectable or potentially resectable ALK-positive NSCLC before neoadjuvant treatment;
13. Cohort 3: Confirmed ALK positive by immunohistochemistry (IHC), fluorescence in situ hybridization (FISH), next-generation sequencing (NGS), or other non-specific sequencing methods before receiving ALK inhibitor therapy;
14. Cohort 3: Signed informed consent form.

Exclusion Criteria:

1. Cohort 1: Patients who have received treatment with Ensartinib after the project has started;
2. Cohort 1: Patients who have received Ensartinib treatment but have not completed the objective efficacy evaluation according to the follow-up cycle specified by the clinical physician;
3. Cohort 1: History of hypersensitivity reactions to active or inactive excipients of Ensartinib or to drugs with similar chemical structures or categories as Ensartinib;
4. Cohort 1: Patients who are participating in other clinical studies outside of this research;
5. Cohort 1: Other circumstances deemed unsuitable for enrollment by the researchers.
6. Cohort 2: Patients who have received Ensartinib treatment before the study started;
7. Cohort 2: Patients who have received other systemic treatments besides Ensartinib;
8. Cohort 2: Neoadjuvant treatment cycles less than 6 weeks or more than 12 weeks;
9. Cohort 2: Patients who have received Ensartinib monotherapy but have not completed the objective efficacy evaluation according to the follow-up cycle specified by the clinical physician;
10. Cohort 2: History of hypersensitivity reactions to active or inactive excipients of Ensartinib or to drugs with similar chemical structures or categories as Ensartinib;
11. Cohort 2: Patients who are participating in other clinical studies outside of this research;
12. Cohort 2: Other circumstances deemed unsuitable for enrollment by the researchers.
13. Cohort 3: Patients who have received neoadjuvant treatment containing Ensartinib but meet the enrollment criteria for Cohort 2;
14. Cohort 3: Patients who have received treatment containing Ensartinib but have not completed the objective efficacy evaluation according to the follow-up cycle specified by the clinical physician;
15. Cohort 3: History of hypersensitivity reactions to active or inactive excipients of Ensartinib or to drugs with similar chemical structures or categories as Ensartinib;
16. Cohort 3: Patients who are participating in other clinical studies outside of this research;
17. Cohort 3: Other circumstances deemed unsuitable for enrollment by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK+
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
MPR | 6month
  Main pathological remission rate

SECONDARY OUTCOMES:
pCR | 6month
  Pathological complete response rate
2-year disease-free survival rate | 2year
  2-year disease-free survival rate
ORR | 1year
  Objective response rate

IPD SHARING:
Plan to Share IPD: No